CLINICAL TRIAL: NCT07187531
Title: A Phase 2b, Randomised, Double-Blind, Placebo-Controlled, Parallel-Arm Dose Finding Study Evaluating the Efficacy and Safety of SAB-142 for Delaying the Progression of Type 1 Diabetes (T1D) in Patients With Stage 3 New Onset of Type 1 Diabetes (NOT1D)
Brief Title: SAFety and Efficacy of Human Anti-thymocyte ImmunoGlobUlin SAB-142 ARresting Progression of Type 1 Diabetes
Acronym: SAFEGUARD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SAb Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SAB-142-201; 2025-521560-36-00 (EU CTIS Number); U1111-1320-2651 (Other: WHO)
Record Dates: First submitted 2025-09-08; First posted 2025-09-23 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- High Dose SAB-142 (Experimental): Part A: Open-label, parallel arm study.
  Part B: Double-blind, placebo-controlled, parallel-arm study. Enrolment into Part B may commence once all participants in Part A have been randomised.
  Interventions: Drug: High Dose SAB-142
- Low Dose SAB-142 (Experimental): Part A: Open-label, parallel arm study.
  Part B: Double-blind, placebo-controlled, parallel-arm study. Enrolment into Part B may commence once all participants in Part A have been randomised.
  Interventions: Drug: Low Dose SAB-142
- Placebo (Placebo Comparator): Part B: This is a double-blind, placebo-controlled, parallel-arm study. Enrolment into Part B may commence once all participants in Part A have been randomised.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: High Dose SAB-142 — High Dose SAB-142
  Arms: High Dose SAB-142
Drug: Low Dose SAB-142 — Low Dose SAB-142
  Arms: Low Dose SAB-142
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a Phase 2b, investigator- and participant-blinded, placebo-controlled, parallel-arm study to evaluate the efficacy, safety and tolerability of SAB 142 in patients with Stage 3 New Onset of Type 1 Diabetes (NOT1D).

ELIGIBILITY:
Inclusion Criteria:

1. Participant and/or appropriate legal guardian must have given written informed consent and/or assent according to local, regional and/or country specific guidance before any study-related activities are carried out and must be able to understand the full nature and purpose of the trial, including possible risks and adverse effects.
2. Males and females 15-40 years old at the time of randomisation in Part A. Males and females 5-40 years old*, inclusive, at the time of randomisation in Part B.
3. Weight ≥16.0 kg at time of randomisation.
4. Participant has received a diagnosis of T1D according to American Diabetes Association criteria within 100 days of randomization. For participants who were initially misdiagnosed with Type 2 diabetes, time from misdiagnosis with Type 2 diabetes to randomization is 100 days. Note: The date of diagnosis is defined as the date of the first insulin dose or any other glucose lowering medication. An extension of no more than 14 days is permitted if a participant has planned and/or is required to receive a vaccination within 30 days prior to randomisation or is completing the 10 day CGM period.
5. Participant has random C-peptide levels of ≥0.2 nmol/L, measured during Screening. One random C-peptide retest during screening period is allowed.
6. Participant completed all scheduled samples for C-peptide collected during the MMTT test during Screening.
7. Participant has a positive result on testing for at least one of the following T1D-related autoantibodies during screening:

   * Glutamic acid decarboxylase 65 (GAD65)
   * Islet antigen 2 (IA-2)
   * Zinc transporter 8 (ZnT8)
   * Insulin autoantibodies (if testing within the first 14 days of insulin treatment)
8. Female participants:

   a. Must be of nonchildbearing potential, i.e., pre-pubertal*, surgically sterilised (hysterectomy, bilateral salpingectomy, bilateral oophorectomy) at least 6 weeks before the screening, or postmenopausal (where postmenopausal is defined as no menses for 12 months without an alternative medical cause and a follicle stimulating hormone (FSH) level consistent with postmenopausal status, per local laboratory guidelines), or b. If of childbearing potential, must: i. Have a negative result on a serum (beta human chorionic gonadotropin [β-HCG]) at screening and a negative urine β-HCG pregnancy test prior to study drug administration on Day 1 of both treatment periods.

   ii. Agree not to become pregnant or donate ova from signing the consent form until the end of study visit.

   iii. If not exclusively in a same-sex relationship or abstinent as a committed lifestyle, must agree to use adequate contraception (which is defined as use of a condom by the male partner combined with use of a highly effective method of contraception from signing the consent and for the duration of the study.

   * Note: Female participants will be considered to be pre-pubertal (and of nonchildbearing potential) if they have not yet started menstruation. This should also be verified by the parent(s)/guardian(s). If a female participant reaches menarche during the study, then she is to be considered as a woman of childbearing potential from that time forwards, and contraceptive requirements will apply.
9. Male participants, if not biologically or surgically sterilised, must:

   1. Agree not to donate sperm from signing the consent form until EOS.
   2. If engaging in sexual intercourse with a female partner who could become pregnant, agree to use adequate contraception (defined as use of a condom combined with use of a highly effective method of contraception from signing the consent form until EOS.
   3. If engaging in sexual intercourse with a female partner who is not of childbearing potential or a same-sex partner, agree to use a condom from signing the consent form until EOS.
10. Prior to receiving study drug, participant must agree to receive locally, regionally and/or country-specific required age-appropriate immunisations. Participants are advised but not required to comply with the guidelines for immunosuppressed individuals and those with chronic disease (diabetes mellitus) according to current local, regional and/or country- specific guidelines. Note: Vaccines are permitted within the timeframes specified in exclusion criterion #17.
11. Participant agrees not to receive other forms of experimental treatment from the time of signing informed consent and for the duration of the study, particularly agents that may be immune modulatory in nature and/or stimulate pancreatic β cell regeneration or insulin secretion.
12. Participant has suitable venous access for blood sampling.
13. Participant is willing and able to comply with all study assessments and adhere to the protocol schedule and restrictions.

Exclusion Criteria:

1. Participant has known allergy, hypersensitivity or moderate to severe allergic reaction including anaphylaxis to natural or recombinant antibodies, biologic treatments, passive vaccines, pork, or any other component of the study drug formulation (including biologic medications).
2. Participant has a known allergy or hypersensitivity to any of the protocol-required concomitant medications.
3. Participant has been an active participant in a therapeutic drug, invasive medical device, or vaccine clinical trial within 12 weeks before Screening Visit (SV)2.
4. Participant has received teplizumab or any investigational immunomodulatory anti-CD3 treatment within any timeframe prior to screening.
5. Participant has a significant uncontrolled renal, cardiac, vascular, pulmonary, gastrointestinal, neurologic, haematologic, rheumatologic, oncologic, psychiatric, or immune deficiency that may interfere with the participant's safely participating in the study or with interpretation of the safety and/or efficacy profile of investigational medicinal product (IMP). For any disorders, a participant with a stable, well-controlled condition that is not felt to interfere with study participation may be enrolled.
6. Participant has any autoimmune disease other than T1D (e.g., latent autoimmune diabetes in adults, rheumatoid arthritis, polyarticular juvenile idiopathic arthritis, psoriatic arthritis, ankylosing spondylitis, multiple sclerosis, systemic lupus erythaematous) that is currently managed with systemic immunotherapy, with the exception of clinically stable thyroid or celiac disease.
7. Participant is prone to infections, or has chronic, recurrent or opportunistic infectious disease, including but not limited to renal, respiratory or skin infections, Pneumocystis carinii, aspergillosis, latent or active granulomatous infection, histoplasmosis, or coccidioidomycosis.
8. Participant has a history of or serologic evidence at screening of current or past infection with human immunodeficiency virus (HIV)-1 or 2, hepatitis B virus (HBV), or hepatitis C virus (HCV) antibodies.
9. Evidence of active or latent tuberculosis (TB) as documented by medical history and examination, chest X-rays (posterior anterior and lateral), and/or TB testing. Note: Blood testing (e.g., QuantiFERON® TB Gold test) is strongly preferred; if not available, any local approved TB test is allowed.
10. Serious systemic viral, bacterial, or fungal infection (e.g., pneumonia, pyelonephritis), infection requiring hospitalization or IV anti-infective treatments or significant acute or chronic viral (including history of recurrent or active herpes zoster, acute or active cytomegalovirus [CMV], Epstein-Barr Virus [EBV] as determined at screening), bacterial, or fungal infection (e.g., osteomyelitis) 30 days before and during screening. Note: Participants with confirmed active EBV or CMV infection based on polymerase chain reaction (PCR) test can be retested; asymptomatic participants with the most recent PCR-negative test are eligible for participation. Participants with an active mild infection at Screening may be enrolled once the symptoms have resolved and all I/E are met. Participants who have an active infection and/or fever ≥38.0°C (100.4°F) within the 48 hours prior to dose administration should not be dosed.
11. Participant has a diagnosis of significant liver disease or at screening ALT and/or AST >2× or total bilirubin of >1.5× of the age- and sex-specific upper limit of normal (ULN) according to the central laboratory and confirmed by repeated tests. Liver function tests can be repeated during screening and if normalised, participant maybe eligible for randomization. Note: Participants with Gilbert's syndrome are allowed to enrol if only total and/or indirect bilirubin are elevated above ULN while ALT, AST, and alkaline phosphatase (ALP) are within the normal laboratory ranges.
12. An individual has any of the following haematologic parameters, confirmed by repeat tests, during Screening:

    * Lymphocyte count: <1000/μL
    * Neutrophil count: <1500/μL
    * Platelet count: <100 000 platelets/μL
    * Haemoglobin: <10 g/dL Note: Specific haematologic, oncologic or other systemic conditions that might otherwise result in exclusion and/or is heretofore unrecognised should be considered in individuals who have one or more blood cell counts below or above the normal ranges.
13. Current or prior (within 5× half-lives before SV2) treatment that is known to cause a significant, ongoing change in the course of T1D or immunologic status, including systemic glucocorticoids, verapamil, baricitinib, and others. Note: Inhaled and topical corticosteroids are allowed. Short courses, i.e., approximately 2 weeks or less, of systemic corticosteroids for transient conditions are allowed.
14. Current or prior (within 5× half-lives before SV2) use of drugs other than insulin to treat hyperglycaemia (e.g., metformin, sulfonylureas, glinides, thiazolidinediones, exenatide, liraglutide, glucagon-like peptide 1 agonists [glucagon-like peptide-1], dipeptidyl peptidase-4 [DPP-IV] inhibitors, or amylin).
15. Current or prior (within 5× half-lives before SV2) use of any medication known to significantly influence glucose tolerance (e.g., atypical antipsychotics, diphenylhydantoin, niacin).
16. Current or planned highly restrictive dietary regimen(s) that would interfere with participant well-being or impact to investigational drug.
17. Recent or planned vaccinations as follows:

    * Live vaccines (e.g., varicella, measles, mumps, rubella, cold-attenuated intranasal influenza vaccine, and smallpox): Within the 30 days before dosing or within 60 days following dosing; or planned/required within 30 days prior to or 60 days following Day 1 of TP2.
    * Recombinant, inactivated or otherwise "non-live" vaccines: Within the 30 days before dosing or within 60 days following dosing; or planned/required within 30 days prior to or 60 days following Day 1 of TP2.
18. Female is lactating and/or plans to lactate with the intent to provide her own breast milk to a baby at any point during the study.
19. An individual who has a history of alcohol, drug, or chemical abuse within 12 months prior to study screening (positive tetrahydrocannabinol is allowed) Note: Abuse is defined according to local, regional and/or country specific guidance. Participants who are tested positive for illicit substances but have a prescription medication to manage their concomitant conditions such as attention-deficit/hyperactivity disorder (ADHD) or others are allowed to participate in the study.
20. An individual who has a medical, psychological or social condition that, in the opinion of the Investigator, would interfere with safe and proper completion of the trial.
21. An individual who is an employee of the Investigator or study site, with direct involvement in the proposed study or other studies under the direction of that Investigator or study site.

Ages: 5 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 159 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Part A: Incidence of treatment-emergent adverse events (TEAEs), adverse events of special interest (AESIs), and serious adverse events (SAEs) | From dose administration through Week 4
Part B: Area under the concentration-time curve (AUC) of C-peptide after a 2 hour mixed meal tolerance test (MMTT) | From dose administration up to Month 12
  This is a measure of endogenous insulin production and β cell function (change from baseline in C-peptide ln [AUC+1] at 12 months)

SECONDARY OUTCOMES:
Part B: Time in tight range (TITR) | At baseline, Months 3, 6, 9 and 12
  Expressed as a daily average of the percentage of time in a 24hour day a participant's glucose is >70 but ≤140 mg/dL (>3.9 to ≤7.8 mmol/L), assessed using continuous glucose monitoring (CGM)
Part B: Haemoglobin A1c (HbA1c) levels | At baseline, Months 3, 6, 9 and 12
  Expressed in % and mmol/mol
Part B: Time in range (TIR) | At baseline, Months 3, 6, 9 and 12
  Expressed as a daily average of the percentage of time in a 24-hour day a participant's CGM reading is >70 but ≤180 mg/dL (>3.9 to ≤10.0 mmol/L), assessed by CGM
Part B: Time above range, assessed by CGM | At baseline, Months 3, 6, 9 and 12
Part B: Time below range, assessed by CGM | At baseline, Months 3, 6, 9 and 12
Part B: Exogenous insulin use | At baseline, Months 3, 6, 9 and 12
  Defined as a daily average in units per kilogram per day (U/kg/day) (total daily insulin based on participant's diary at predefined study periods)
Part B: Number of clinically important episodes | At baseline, Months 3, 6, 9 and 12
  Defined as the total number of Level 2 and 3 hypoglycaemic events and/or episodes of cognitive impairment requiring external assistance for recovery (participant's diary and CGM-based)
Part B: Proportion of participants with partial clinical remission | At baseline, Months 3, 6, 9 and 12
  Defined as an insulin requirement of <0.25 units per kg of body weight per day and HbA1c <6.5% (47 mmol/mol)
Part B: Proportion of participants with partial remission | At baseline, Months 3, 6, 9 and 12
  Defined as insulin-dose adjusted A1c (IDAA1c) + [4 × insulin dose (units per kilogram per 24 h) ≤9
Part B: Total BETA-2 score, comprised of fasting plasma glucose (mmol/L), HbA1c (%), daily insulin (U/kg), and fasting C-peptide (nmol/L) | At baseline, Months 3, 6, and 12
Part B: Insulin dose-adjusted A1c (IDAA1C) | At baseline, Months 3, 6, 9 and 12
Part B: Incidence of TEAEs, AESIs, and SAEs | From dose administration through Month 12
Part B: SAB-142 serum concentrations | Days 1 and 2 of each treatment period (pre- and post- dose/end of infusion [EOI]), plus Weeks 1, 4, and Months 3, 6, and 7
Part B: Incidence of anti-SAB-142 antibodies including optional neutralising antibodies (nAbs) in serum | At baseline, Week 4, Months 3, 6, 7, 9 and 12
Part B: Titres of anti-SAB-142 antibodies including optional neutralising antibodies (nAbs) in serum | At baseline, Week 4, Months 3, 6, 7, 9 and 12
Part B: Immunophenotyping (IPT) | At baseline (Day 1, pre-dose), Week 4, Months 3, 6, 7, 9 and 12

CONTACTS AND LOCATIONS:
Locations (65):
- United States (17):
  - University of California San Francisco Benioff Children's Hospital, San Francisco, California
  - University of Colorado - Barbara Davis Center for Diabetes, Aurora, Colorado
  - University of Florida College of Medicine, Gainesville, Florida
  - University of Miami - Gables One Tower, Miami, Florida
  - Children's Healthcare of Atlanta (CHOA) - Center for Advanced Pediatrics, Atlanta, Georgia
  - IUH - Riley Hospital for Children - Riley Outpatient Center - Pediatric Diabetes & Endocrinology, Indianapolis, Indiana
  - Harvard Medical School - Joslin Diabetes Center and Joslin Clinical (JDS), Boston, Massachusetts
  - Children's Mercy Hospital Kansas - Pediatric Care Clinic, Kansas City, Missouri
  - University at Buffalo MD Physicians Group, Buffalo, New York
  - N.C. Children's Hospital - Children's Specialty Clinics - Chapel Hill at Carolina Pointe II, Chapel Hill, North Carolina
  - Sanford Medical Center Fargo, Fargo, North Dakota
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Cook Children's Medical Center, Fort Worth, Texas
  - Texas Children's Hospital - Clinical Care Center - Pediatric Renal Clinic, Houston, Texas
  - University of Virginia Health System - Pediatric Diabetes Clinic, Charlottesville, Virginia
  - Benaroya Research Institute at Virginia Mason, Seattle, Washington
  - Mary Bridge Children's Outpatient Center - Tacoma, Tacoma, Washington
- Australia (6):
  - Queensland Children's Hospital, Brisbane
  - Government of Western Australia - Child and Adolescent Health Service - Perth Children's Hospital, Nedlands
  - The Royal Children's Hospital Melbourne, Parkville
  - The Royal Melbourne Hospital (RMH), Parkville
  - Royal North Shore Hospital (RNSH), St Leonards
  - Westmead Hospital, Westmead
- Austria (4):
  - Medizinische Universitaet Graz - Klinik fuer Innere Medizin, Graz
  - Medizinische Universität Innsbruck, Innsbruck
  - Medizinische Universitaet Graz - Universitaetsklinik fuer Kinder und Jugendheilkunde, Vienna
  - Medizinische Universitaet Wien - Universitaetsklinik fuer Kinder und Jugendheilkunde, Vienna
- Belgium (3):
  - Universitair Ziekenhuis Brussel, Jette
  - UZ Leuven, Leuven
  - Groupe sante CHC - Clinique du MontLegia, Liège
- Steno Diabetes Center, Herlev, Denmark
- Finland (2):
  - Helsingin Yliopistollinen Keskussairaala, Helsinki
  - Turun Yliopistollinen Keskussairaala (TYKS), Turku
- France (2):
  - Universite Paris Descartes - Institut Cochin, Paris
  - Assistance Publique-Hopitaux de Paris (AP-HP) - Hopital Universitaire Robert-Debre, Paris
- Germany (3):
  - Klinikum Augsburg, Augsburg
  - Hannoversche Kinderheilanstalt, Hanover
  - Technische Universität Munich, Oberschleißheim
- Italy (3):
  - IRCCS Ospedale San Raffaele, Milan
  - Azienda Ospedaliero Universitaria Maggiore della Carità di Novara, Turin
  - Azienda Ospedaliera Universitaria Integrata Verona-Ospedale della Donna e del Bambino_Borgo Trento, Verona
- Hospital of Lithuanian University of Health Sciences Kauno Klinikos, Kaunas, Lithuania
- New Zealand (6):
  - Waitemata District Health Board- North Shore Hospital, Auckland
  - Aotearoa Clinical Trials, Auckland
  - New Zealand Clinical Research - Christchurch, Christchurch
  - Dunedin Hospital, Dunedin
  - Waikato Hospital, Hamilton
  - Wellington Regional Hospital, Wellington
- Poland (5):
  - Uniwersytecki Szital Klniczny w Opolu, Opole
  - SZPITAL KLINICZNY im. Karola Jonschera - UNIWERSYTETU MEDYCZNEGO im. Karola Marcinkowskiego, Poznan
  - Warszawski Uniwersytet Medyczny - Klinika Pediatrii, Warsaw
  - Instytut Diabetologii, Warsaw
  - MTZ Clinical Research Sp. z o.o., Warsaw
- University Children's Hospital Ljubljana (UCHL), Ljubljana, Slovenia
- Spain (3):
  - Hospital de Cruces, Barakaldo
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen Macarena, Seville
- United Kingdom (8):
  - Cambridge University Hospitals NHS Foundation Trust - Addenbrookes Hospital, Cambridge
  - Noahs Ark Childrens Hospital for Wales, Cardiff
  - NHS Lothian - Royal Hospital for Sick Children, Edinburgh
  - Alder Hey Children's NHS Foundation Trust, Liverpool
  - Barts Health NHS Trust - The Royal London Hospital, London
  - University College London Hospitals NHS Foundation Trust - University College Hospital, London
  - Nottingham University Hospitals NHS Trust - Queen's Medical Centre (QMC), Nottingham
  - Oxford University Hospitals NHS Trust - John Radcliffe Hospital, Oxford